CLINICAL TRIAL: NCT04297904
Title: Associations Between Urinary Incontinence, Sedentary Behaviour and Other Health-related Outcomes in Nursing Homes in Catalonia: the OsoNaH Project
Brief Title: Urinary Incontinence and Sedentary Behaviour in Nursing Homes
Acronym: OsoNaH
Status: Completed | Type: Observational
Sponsor: University of Vic - Central University of Catalonia (Other)
Collaborators: Glasgow Caledonian University (Other); University Ramon Llull (Other); Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Javier Jerez Roig, Ph.D. Research Delegate of the Faculty of Health Sciences and Wellfare of University of Vic - Central University of Catalonia. Head of research group on Methodology, Methods, Models and Outcomes of Health and Social Science (M3O), University of Vic - Central University of Catalonia
Other Study IDs: ONH001
Record Dates: First submitted 2020-02-28; First posted 2020-03-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Urinary Incontinence in Old Age; Sedentary Behavior
Keywords: Nursing home; Older people; Urinary incontinence; Sedentary behaviour; Functioning
MeSH Terms: conditions — Sedentary Behavior; Urinary Incontinence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Sedentary behaviour — To assess sedentary behaviour each participant will wear an activity monitor (PAL Technologies, Scotland). The resident will wear the monitor on their right thigh for 24 hours per day over seven days continuously.
Diagnostic Test: Urinary Incontinence — The presence of IU, assessed by the Minimum Data Set (MDS) version 3.0, and used together with the International Consultation on Incontinence Questionnaire-Short Form to characterize the incontinence.

SUMMARY:
The increase of the older adult population in the past years has generated an important impact on chronic conditions and geriatric syndromes like dementia, falls and urinary incontinence (UI). To better understand IU seems warranted because of its socioeconomic and health impact. Nursing home (NH) residents are the frailest segment of our population, with very low physical activity levels and highly sedentary. Several studies had shown that physical activity levels and time and patterns of sedentary behaviour (SB) are independent risk factors for many health issues. As far as the investigators know, there is no evidence supporting the relation between IU and SB, and no information about the incidence of IU in NH residents living in Catalonia (Spain).

This project consists of two stages: stage 1 will conduct a cross-sectional study using mixed methodology (qualitative and quantitative), and a 2-year longitudinal study (stage 2). Stage 1 has the main objective of verifying the prevalence of IU and its associated factors in NH residents in Barcelona (Spain), as well as analyse the association between IU (and their types) with SB time and patterns. In addition, the proportion of geriatric residents who receive control measures for their IU, and whether they receive SB-related interventions from health professionals of the institution will be also explored. Finally, the investigators aim to understand the experience of NH residents and the health professionals who care for them about the characteristics, burden and barriers of having IU. Stage 2 has the main objective to verify the incidence of the functional and continence decline, falls, hospitalizations and mortality, as well as their predictive factors in older care/nursing home residents in Barcelona (Spain). Specific objetives are to assess the evolution of each activity of daily living and the causes of hospitalization and death in geriatrics residents for a period of 2 years and to verify the incidence of recurrent falls (one or more falls), and analyse the consequences of falls (fractures, hospitalizations, among others) among the residents. Potential risk and protective factors for mortality due to COVID-19 and its impact on functioning and hospitalizations will also be analyzed. Finally, the stage 2 of the project aims at creating a specific instrument for the evaluation of frailty in institutionalized older people, based on the main predictive factors of functional decline.

DETAILED DESCRIPTION:
The low birth rate and an increased life expectancy are transforming the age pyramid of the European Union (EU); probably the most important change will be the marked transition towards an aged society, a characteristic that is already evident in several EU member states. In 2017, the 65+ older adult's population had an increase of 0.3% compared to the previous year, and an increase of 2.4% compared to the previous 10 years. People over 80 years old are increasing at a faster rate than any other age segment of the EU population. This increase is probably linked to a growing demand for long-term care, which represents a significant overload on public health resources. Care/nursing homes are the main providers of long-term care. One of four older adults will spend a period of their life in a care/nursing home, and the dependence for such care will persist until their dead. The older adults who live in a nursing home are the most fragile of our society with high levels of physical dependence and one third of them suffering from cognitive impairment. An acute hospitalization typically is associated with multiple diseases in older people, and disability is frequently followed by high rates of progressive physical decline and mortality in the years following discharge. It is well known that hospital admission can change normal aging due to adverse health outcomes after hospitalization, especially in terms of functional decline, mortality frailty and cognitive impairment.

Frailty is one of the most important concerns regarding our aging population. Evidence grows that the syndrome is linked to several important health outcomes, prevalent in all countries and is a leading contributor to functional decline and early mortality in older adults. The last consensus defined frailty as "a clinical state in which there is an increase in an individual's vulnerability for developing an increased dependency and/or mortality when exposed to a stressor".

The decline in functionality is one of the main issues that affects older people because it limits their autonomy and leads to dependency. In older people, functional capacity can be defined as the ability to carry out a set of activities necessary for an independent life, the ability to carry out basic activities of daily living (BADL), those related to self-care and survival (such as bathing and eating), and more complex actions called instrumental activities (such as shopping and transportation). Functionality decline lead to high financial costs and are close associated with frailty, mobility problems, and increased risk of falls, dependency, hospitalization, and death. The association between functional decay and urinary incontinence (UI) could be bidirectional, which can lead to a cycle where continence reduction results in functional decline, and functional decline leads to further decrease in urinary continence.

The prevalence of UI in Spain is approximately 10% in women between 25 and 64 years old and over 50% in those over 65 years old. In the domain of nursing homes, this proportion is around 50% and is frequently associated with cognitive impairment, physical inactivity and immobility syndrome, among other factors. In this context, we can find a type of UI described as "functional" that it's caused by the inability to move to the bathroom independently, due to a physical or cognitive problem (e.g. dementia). Most older adults mistakenly believe that incontinence is part of the normal aging process and / or is an irresolvable problem. However, UI is a geriatric syndrome that represents an indicator of frailty and quality of health care, as well as a risk factor for pressure ulcers, falls, fractures and even urinary sepsis or death.

Falls, though preventable, are common among older adults, and the resulting injuries can threaten their health, independence, and lives. In 2014, 30% of older adults (aged > 65 years) in the United States reported falling at least once, and the estimated 29 million falls that year resulted in 7 million injuries and approximately 27,000 deaths. The evidence and research in Spain, shows that 30% of people over 65, independent and autonomous will be affected by an annual fall. This percentage increases progressively as age increases, because age is one of the main factors of risk in falls, being older people the ones with highest risk of suffering injuries, increased dependence, disabilities, institutionalization in centers and death, considering itself as a factor of frailty. In people over 75 years old its risk of fall rises to 35%, and in people over 80 years old it reaches 50%. Several studies estimate that this prevalence increases up to 50% in the case of institutionalized older people. Falls are an important public health problem, being an underdiagnosed problem, because when there are no physical consequences, do not usually go to the health system.

Previous investigations followed by decades of research, confirm that nursing home residents are the less physically active and spend most of their awake time inactives). Doing regular physical activity (PA) limit the development and progression of most prevalent chronic diseases. However, time spent in SB has increased considerably in the last three decades and increases with age. SB has been gaining recognition as a risk factor of specific health conditions and reduced mobility, sometimes independent of PA levels. A typical day for a resident will consist in a sequence of periods of SB, light intensity PA (LPA) and moderate to vigorous intensity PA (MVPA). Care/nursing home residents spend an average of 79% of their day sedentary, 20% in LPA and 1% in MVPA.

Regarding the association between SB and the UI, there is little evidence available. In a recent literature review on the association between SB and UI in women, the review concluded that information available was limited, although suggested that SB could be considered a risk factor for UI in women. If we review the little existing literature concerning the association between SB and UI, there is a consensus among the authors on low levels of PA and prolonged patterns of SB could be direct risk factors for UI in older adults or in the older women, and there is a lack of complementary studies of higher quality in the association between SB and UI.

On the other hand, the COVID-19 pandemic has emerged as a new major public health issue especially affecting NHs. This virus has been shown to be particularly deadly for older adults and those with certain underlying medical conditions. In relation to deaths from COVID-19 in Spain, 87% of the reported deaths were 70 years or more and a 95% presented comorbidity. The population living in NH, generally with older age and multiple comorbidities, are the most vulnerable to COVID-19. In Catalonian NHs 28,418 suspected cases, 11,560 confirmed positive cases and 3,055 deaths were reported until May 2020. Due to the vulnerability of NHs themselves to outbreaks of respiratory diseases and the frailty of NH population, there is a need of analysing the impact of COVID-19 in NH residents in terms of mortality, hospitalisation, as well as other health, social and cognitive-related variables. We also want to learn about the potential risk and protective factors for mortality due to COVID-19 and the impact of this disease on funtioning and hospitalizations.

For all the reasons cited above, they lead us to think that there is a gap in the description of nursing home residents. Consequently, the stage 1 of this study aims at knowing the current state of health-related outcomes of nursing home older adults and the factors that influence their quality of life. Reducing SB patterns and ensuring an increase in PA in an individualized and progressive way can contribute to the stabilization of chronic cardio metabolic pathologies, improve their muscular quality and cardiopulmonary capacity, improve their biopsychosocial sphere and promote their socialization with other residents and health professionals and finally increase their participation in the nursing home. However, the certain association between SB and UI remains unclear. The OsoNaH project will try to cover this lack of knowledge and define the possible aetiology and associated factors with the different types of UI and SB, in order to determine new ways of intervention, treatment and care for the nursing home residents. Finally the stage 2 aims to better know the characteristics of functional decline, continence decline, falls, hospitalizations and mortality due to the importance and impact they generate on older people and their caregivers. This project may help to develop of new lines of interventions, management and treatment. Also, this study will try to fill de gap of knowledge in the region of Central Catalonia about this issues. So it is considered necessary to know from an interdisciplinary and longitudinal field, the evolution / appearance and predictive factors of functional decline, continence decline, falls, hospitalizations and mortality of institutionalized older people.

ELIGIBILITY:
Inclusion Criteria for the quantitative part:

* All nursing home residents (male or female) 65 years of age or older who live in the institution permanently who voluntary will to participate in the study.

Exclusion Criteria for the quantitative part: :

* Subjects in coma or palliative care (prognosis of short life).

Inclusion criteria for the qualitative part (residents):

* Voluntary participation in the study.
* Be diagnosed with UI for at least 6 months
* Be able to express themselves verbally.

Inclusion criteria for the qualitative part (professionals):

* Voluntary participation in the study
* Caring for older people with UI for at least 6 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: All nursing home residents, both sexes, 65 years of age or older who live in the institution permanently willing to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Urinary Incontinence | January 2020 to July 2020 (cross-sectional)
  The presence of IU assessed by the Minimum Data Set (MDS) version 3.0
Patterns of sedentary behaviour | January 2020 to July 2020 (cross-sectional)
  Patterns of sedentary behaviour (SB) with monitors (PAL Technologies, Scotland).
Functional decline | January 2020 to March 2022 (longitudinal, follow-up)
  Modified (Likert 5-point scale) Barthel Index, assessed every 6 months
Continence decline | January 2020 to march 2022 (longitudinal, follow-up)
  Minimum Data Set (MDS) version 3.0, assessed every 6 months
Incidence of falls | January 2020 to March 2022 (longitudinal, follow-up)
  Prospective register of falls (date, place and consequence/s)
Hospitalizations | January 2020 to March 2022 (longitudinal, follow-up)
  Prospective register of hospitalizations (date and cause)
Mortality | January 2020 to March 2022 (longitudinal, follow-up)
  Prospective register of deaths (date and cause)

SECONDARY OUTCOMES:
Sociodemographic variables | January 2020 to July 2020
  Sociodemographic variables (sex, age, civil status, education level, type of institution (public versus private / concerted) and time of residence in the institution.)
Lower urinary tract symptoms | January 2020 to July 2020
  Number and proportion of participants with lower urinary tract symptoms with the International Prostate Symptoms Score and urinary infection for the last 30 days.
Faecal incontinence | January 2020 to July 2020
  Faecal incontinence according to Minimum Data Set version 3.0 (MDS 3.0)
Intake of liquids and diuretic drinks | January 2020 to July 2020
  Diary
Handgrip strength | January 2020 to July 2020
  Dynamometer (2 trials per hand)
Physical performance | January 2020 to July 2020
  Short Physical Performance Battery (SPPB)
Mobility | January 2020 to July 2020
  Rivermead Mobility Index
Frailty | January 2020 to July 2020
  Clinical Frailty Scale
Basic activities of daily living | January 2020 to July 2020
  Modified (Likert 5-point scale) Barthel Index
Physical activity programs | January 2020 to July 2020
  What kind of physical activity programme, the frequency of the sessions weekly, the dose of exercise of each session, the duration of the whole session, who provides the session, where the session is performed and if the session is individually or in group).
Incontinence programs | January 2020 to July 2020
  What kind of programs are being applied to control and treat urinary and faecal incontinence in nursing homes
Medication intake | January 2020 to July 2020
  According to the Anatomical Therapeutic Chemical classification system and the Defined Daily Dose (ATC/DDD)
Health conditions | January 2020 to July 2020
  Number and proportion of participants with chronic diseases, delirium and pressure ulcers
Toxic habits | January 2020 to July 2020
  Number and proportion of participants who have smoked ever and are taking alcohol currently
Cognitive status | January 2020 to July 2020
  Pfeiffer Scale, with final score ranging from 0 (normal) to 10 (total cognitive impairment)
Depressive symptoms | January 2020 to July 2020
  15-item Yesavage Geriatric Depression Scale, with final score ranging from 0 (normal) to 15 (severe depression)
Anxiety | January 2020 to July 2020
  Hospital Anxiety and Depression Scale (HADS), with final score ranging from 0 (normal) to 21 (severe anxiety)
Number births | January 2020 to July 2020
  Using the NH register
Type of births | January 2020 to July 2020
  Using the NH register
Number of falls | January 2020 to July 2020
  During the last year, according to the NH register
Nutritional status | January 2020 to July 2020
  Mini Nutritional Assessment Test, ranging from 0 (malnutrition) to 30 (normal)
Biochemical evaluation | January 2020 to July 2020
  Amount of Vitamin D, albumin and pre-albumin, PCR (Protein C-Reactive) extracted from the routine analysis of the residents.
Body composition | January 2020 to July 2020
  Percentage (%) of body fat, % of fat-free mass and % of body water assessed by a Tanita TBF-300 bioimpedance device
Social network | January 2020 to July 2020
  Lubben Social Network Scale ranging from 0 to 30, with a higher score indicating more social engagement.
Loneliness | January 2020 to July 2020
  6-item Gierveld Loneliness Scale ranging from 0 (not lonely) to 6
COVID-19 | June 2020 to March 2022 (longitudinal, follow-up)
  Date and result of diagnosis test/s for COVID-19 (PCR or serological antibody test)
Suspected case of COVID-19 | June 2020 to March 2022 (longitudinal, follow-up)
  In the previous 6 months, the resident had symptoms compatible with COVID-19 (cough, fever and/or breathing difficulties) without COVID-19 diagnosis test confirmation
Frailty | June 2020 to March 2022 (longitudinal, follow-up)
  Level of resident's frailty assessed with the Clinical Frailty Scale
Change in medication | June 2020 to March 2022 (longitudinal, follow-up)
  Any change in the regular medication in the last 6 months (include the name of the med, dose and the duration of treatment)
Quality of life (European Quality of Life-5 Dimensions) | January 2020 to July 2020
  final score for Spain ranges between 1 (full health) to -0.654 (worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Minobes Molina, PhD, Principal Investigator — M3O; Javier Jerez-Roig, PhD, Professor, Principal Investigator — M3O
Locations (15):
- Spain (15):
  - Residència Sant Gabriel. Nursing home, Centelles, Barcelona
  - Casal Oller. Nursing home, els Hostalets de Balenyà, Barcelona
  - Casal de la Santa Creu. Nursing home, L'Esquirol, Barcelona
  - Residència Cantonigròs. Nursing home, L'Esquirol, Barcelona
  - Residència Aura. Nursing home, Manlleu, Barcelona
  - Residència els Tells. Nursing home, Montesquiu, Barcelona
  - Els Munts. Nursing home, Sant Boi de Lluçanès, Barcelona
  - Fundació Gallifa. Nursing home, Sant Hipòlit de Voltregà, Barcelona
  - Els Bons Amics. Nursing home, Seva, Barcelona
  - Hotel Residència el Prat. Nursing home, Tona, Barcelona
  - Residència Prudenci. Nursing home, Tona, Barcelona
  - Residencia Rocapravera. Nursing home, Torelló, Barcelona
  - Funcació Privada de Gestió Clear - Residència Centre de Dia SAITS. Nursing home, Vic, Barcelona
  - Residencia el Nadal. Nursing home, Vic, Barcelona
  - University of Vic - Central University of Catalonia. Facultat de Ciències de la Salut i el Benestar; Afiliation with the M3O research group, Vic, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Escriba-Salvans A, Rierola-Fochs S, Farres-Godayol P, Molas-Tuneu M, de Souza DLB, Skelton DA, Goutan-Roura E, Minobes-Molina E, Jerez-Roig J. Risk factors for developing symptomatic COVID-19 in older residents of nursing homes: A hypothesis-generating observational study. J Frailty Sarcopenia Falls. 2023 Jun 1;8(2):74-82. doi: 10.22540/JFSF-08-074. eCollection 2023 Jun. PMID 37275659
- [Derived] Farres-Godayol P, Jerez-Roig J, Minobes-Molina E, Yildirim M, Goutan-Roura E, Coll-Planas L, Escriba-Salvans A, Molas-Tuneu M, Moreno-Martin P, Rierola-Fochs S, Rierola-Colomer S, Romero-Mas M, Torres-Moreno M, Naudo-Molist J, Bezerra de Souza DL, Booth J, Skelton DA, Gine-Garriga M. Urinary incontinence and sedentary behaviour in nursing home residents in Osona, Catalonia: protocol for the OsoNaH project, a multicentre observational study. BMJ Open. 2021 Apr 20;11(4):e041152. doi: 10.1136/bmjopen-2020-041152. PMID 33879481